CLINICAL TRIAL: NCT02279862
Title: A Phase 2, Randomized, Double-Blind Study of Ipilimumab Administered at 3 mg/kg vs 10 mg/kg in Adult Subjects With Metastatic Chemotherapy-Naïve Castration Resistant Prostate Cancer Who Are Asymptomatic or Minimally Symptomatic
Brief Title: Safety and Efficacy Study of Ipilimumab 3 mg/kg Versus Ipilimumab 10 mg/kg in Subjects With Metastatic Castration Resistant Prostate Cancer Who Are Chemotherapy Naive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-437; 2014-002987-34 (EudraCT Number)
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Ipilimumab 3 mg/kg (Experimental): Ipilimumab 3 mg/kg injection intravenously every 3 weeks for 4 doses in Induction phase. Subjects that are eligible to receive Ipilimumab in the Maintenance phase will be dosed every 12 weeks for a maximum of 3 years since the first induction dose
  Interventions: Drug: Ipilimumab
- Arm 2: Ipilimumab 10 mg/kg (Experimental): Ipilimumab 10 mg/kg injection intravenously every 3 weeks for 4 doses in Induction phase. Subjects that are eligible to receive Ipilimumab in the Maintenance phase will be dosed every 12 weeks for a maximum of 3 years since the first induction dose
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: Yervoy™

SUMMARY:
The purpose of this study is to examine the safety and effectiveness (how well the drug works) of two different doses (3 mg/kg and 10 mg/kg) of Ipilimumab (Yervoy™) in patients with metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
Prostate Cancer Clinical Trials Working Group 2 (PCWG2)

Response Evaluation Criteria In Solid Tumors (RECIST)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Prostate cancer with metastases
* Prostate cancer should be castration resistant
* Progression during hormonal therapy

Exclusion Criteria:

* Visceral metastases (eg liver, lung or brain metastases)
* Prior treatment with any immunotherapy for prostate cancer
* Prior or ongoing cytotoxic therapy for prostate cancer
* Autoimmune disease
* Inadequate hematologic, renal, or hepatic function

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (43):
- United States (11):
  - San Francisco Oncology Associates, San Francisco, California
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Baptist Cancer Institute, Jacksonville, Florida
  - Cancer Center Of Kansas, Wichita, Kansas
  - North Mississippi Med Center, Tupelo, Mississippi
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Providence Portland Medical Center, Portland, Oregon
  - Northwest Cancer Specialists, Pc, Tualatin, Oregon
  - University of Pittsburgh Cancer Institute Cancer Services, Pittsburgh, Pennsylvania
  - Texas Oncology, Houston, Texas
  - Virginia Cancer Institute, Richmond, Virginia
- Australia (3):
  - Local Institution, St Leonards, New South Wales
  - Local Institution, Wahroonga, New South Wales
  - Local Institution, Parkville, Victoria
- Chile (3):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Recoleta, Santiago de Chile
  - Local Institution, Santiago, Santiago Metropolitan
- France (6):
  - Local Institution, Clermont-Ferrand
  - Local Institution, Marseille
  - Local Institution, Poitiers
  - Local Institution, Rennes
  - Local Institution, Saint-Herblain
  - Local Institution, Villejuif
- Germany (10):
  - Universitaetsklinikum Aachen, Aachen
  - Uniklinik Heidelberg, Heidelberg
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Magdeburg, Magdeburg
  - Universitaetsklinikum Mannheim, Mannheim
  - Local Institution, Marktredwitz
  - Klinikum rechts der Isar der TU, München
  - Urologische Praxis, Rostock
  - Urologische Gemeinschaftspraxis Dres Stammel U. Garcia, Wesel
  - Dgu Urologie, Wuppertal
- Italy (2):
  - Local Institution, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
- Local Institution, Amsterdam, Netherlands
- Spain (4):
  - Local Institution, Barcelona
  - Local Institution, Hospitalet de Llobregat - Barcelona
  - Local Institution, Seville
  - Local Institution, Valencia
- United Kingdom (3):
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Guildford, Surrey

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 82 participants were enrolled; 53 were randomized; 51 were treated with study drug. 29 were not randomized due to screening failures. 2 were randomized and not treated due to administrative reason by sponsor and "other" reason
Groups:
- Ipilimumab 3 mg/kg: Ipilimumab at 3 mg/kg was administered by intravenous (IV) infusion over a time period of 60-100 minutes, based on body weight. Induction Phase dosing consisted of a single dose every 3 weeks (Q3W) for 4 doses. This was followed by Maintenance Phase dosing of a single dose every 12 weeks (Q12W). Treatment was for a maximum treatment period of 3 years from the first induction dose of blinded study therapy, or until subject met treatment stopping criteria.
- Ipilimumab 10 mg/kg: Ipilimumab at 10 mg/kg was administered by intravenous (IV) infusion over a time period of 60-100 minutes, based on body weight. Induction Phase dosing consisted of a single dose every 3 weeks (Q3W) for 4 doses. This was followed by Maintenance Phase dosing of a single dose every 12 weeks (Q12W). Treatment was for a maximum treatment period of 3 years from the first induction dose of blinded study therapy, or until subject met treatment stopping criteria.
Period: Overall Study
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Started | 26 | 27
Treated | 25 | 26
Completed | 0 (Completed treatment in induction period) | 2 (Completed treatment in induction period)
Not Completed | 26 | 25
Not completed — Study drug toxicity | 3 | 6
Not completed — No longer meets criteria | 0 | 1
Not completed — Administrative reason by sponsor | 0 | 1
Not completed — Disease progression | 5 | 2
Not completed — Study closed by sponsor | 16 | 13
Not completed — Other | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Median (Full Range); unit: years] | 66.00 (8.23) [50.00 to 85.00] | 66.50 (9.98) [49.00 to 87.00] | 66.00 (9.08) [49.00 to 87.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 26 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Experienced Immune-related Adverse Events (irAEs)
Description: The total number of participants with immune-related adverse events of any grade is reported for each arm.
Time Frame: From first dose of ipilimumab to last dose plus 90 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 25 | 26
Participants | 13 | 18

2. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: rPFS was defined as the time from the date of randomization until the date of disease progression based on radiographic evidence and/or death from any cause, whichever occurs first. Radiographic disease progression is defined as: Confirmed bone disease progression according to criteria adapted from the Prostate Cancer Clinical Trials Working Group 2 (PCWG2), OR Non-bone disease progression according to the modified Response Evaluation Criteria In Solid Tumors (RECIST) 1.1. After termination of the study, collection of tumor assessments and other data to support the efficacy analyses was no longer required in patients who discontinued study treatment. As a result, the presented efficacy results are based on limited data. The number of participants with reported radiographic progression is shown.
Time Frame: From date of randomization until disease progression or death (assessed up to December 2016, approximately 24 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 26 | 27
Participants | 4 | 3

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death. For those participants who have not died, OS was censored at the last date the participant was known to be alive. After termination of the study, collection of tumor assessments and other data to support the efficacy analyses was no longer required in patients who discontinued study treatment. As a result, the presented efficacy results are based on limited data. The total number of reported deaths is shown.
Time Frame: From randomization to death from any cause (assessed up to December 2016, approximately 24 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 26 | 27
Participants | 4 | 6

4. Secondary Outcome: Prostate Specific Antigen Progression-free Survival (PSA PFS)
Description: Prostate specific antigen progression-free survival (PSA PFS) was defined as the time from randomization to the earliest date of PSA progression or death, whichever occurs earlier. Participants who did not progress or die were censored at the last PSA assessment date. After termination of the study, collection of tumor assessments and other data to support the efficacy analyses was no longer required in patients who discontinued study treatment. As a result, the presented efficacy results are based on limited data. The number of participants with reported PSA progression is shown.
Time Frame: From randomization to the earliest date of PSA progression or death, whichever comes earlier (assessed up to December 2016, approximately 24 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 26 | 27
Participants | 4 | 3

5. Secondary Outcome: Time to Pain Progression
Description: Pain progression was defined as an increase in BPI-SF pain Item #3 score of >= 2 point from baseline maintained over 2 consecutive periods. After termination of the study, collection of tumor assessments and other data to support the efficacy analyses was no longer required in patients who discontinued study treatment, and presented efficacy results are based on limited data. The number of participants with reported pain progression is shown.
Time Frame: From randomization until pain progression (assessed up to December 2016, approximately 24 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 26 | 27
Participants | 0 | 1

6. Secondary Outcome: Prostate Specific Antigen Response Rate
Description: PSA response rate was defined as the proportion of participants with a 50% or greater decrease from baseline to the lowest post-baseline PSA result (confirmed 3 weeks later) for each randomized arm. After termination of the study, collection of tumor assessments and other data to support the efficacy analyses was no longer required in patients who discontinued study treatment. As a result, the presented efficacy results are based on limited data. The number of participants showing PSA response is shown.
Time Frame: From baseline to PSA response (assessed up to December 2016, approximately 48 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab 3 mg/kg | Ipilimumab 10 mg/kg
Number analyzed (Participants) | 26 | 27
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From date of first dose to date of last dose of study therapy plus 90 days
Groups:
- 10 MG/KG IPILIMUMAB: Ipilimumab at 10 mg/kg was administered by intravenous (IV) infusion over a time period of 60-100 minutes, based on body weight. Induction Phase dosing consisted of a single dose every 3 weeks (Q3W) for 4 doses. This was followed by Maintenance Phase dosing of a single dose every 12 weeks (Q12W). Treatment was for a maximum treatment period of 3 years from the first induction dose of blinded study therapy, or until subject met treatment stopping criteria.
- 3 MG/KG IPILIMUMAB: Ipilimumab at 3 mg/kg was administered by intravenous (IV) infusion over a time period of 60-100 minutes, based on body weight. Induction Phase dosing consisted of a single dose every 3 weeks (Q3W) for 4 doses. This was followed by Maintenance Phase dosing of a single dose every 12 weeks (Q12W). Treatment was for a maximum treatment period of 3 years from the first induction dose of blinded study therapy, or until subject met treatment stopping criteria.
Arm/Group | 10 MG/KG IPILIMUMAB | 3 MG/KG IPILIMUMAB
Serious Adverse Events (participants affected / at risk) | 15/26 | 6/25
Other Adverse Events (participants affected / at risk) | 22/26 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG IPILIMUMAB (N=26) | 3 MG/KG IPILIMUMAB (N=25)
Myocardial infarction (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG IPILIMUMAB (N=26) | 3 MG/KG IPILIMUMAB (N=25)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Colitis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 12 | 10
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Fatigue (General disorders) | 9 | 4
Mucosal inflammation (General disorders) | 2 | 0
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 6 | 3
Conjunctivitis (Infections and infestations) | 0 | 2
Systemic infection (Infections and infestations) | 0 | 2
Weight decreased (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Nocturia (Renal and urinary disorders) | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 9 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 4

LIMITATIONS AND CAVEATS:
After termination of the study, collection of tumor assessments and other data to support the efficacy analyses was no longer required in patients who discontinued study treatment. As a result, the presented efficacy results are based on limited data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.